CLINICAL TRIAL: NCT05673811
Title: A Phase IIb, Open-label, Randomized Study of Nab-Paclitaxel and Gemcitabine and Plus/Minus VCN-01 in Patients With Metastatic Pancreatic Cancer
Brief Title: Study of Nab-Paclitaxel and Gemcitabine and Plus/Minus VCN-01 in Patients With Metastatic Pancreatic Cancer
Acronym: VIRAGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theriva Biologics SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-VCNA-003
Record Dates: First submitted 2022-11-03; First posted 2023-01-06 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Adenocarcinoma; Metastatic
Keywords: Cancer; Pancreatic adenocarcinoma; metastatic; oncolytic virus; VCN-01; Gemcitabine; Nab-Paclitaxel
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1-SoC (Active Comparator): Nab-paclitaxel and gemcitabine as SoC.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine
- Arm 2 -VCN-01 + SoC (Experimental): A maximum of two (2) doses of VCN-01 administrated as a single IV infusion in combination with nab-paclitaxel and gemcitabine as SoC.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Genetic: VCN-01

INTERVENTIONS:
Drug: Nab-paclitaxel — Nab-paclitaxel administered as an IV infusion at a rate of 125 mg/m2. Nab-paclitaxel is administered on Day 1, Day 8 and Day 15 of each 28-day cycles.
Drug: Gemcitabine — Gemcitabine administered as an IV infusion at a dose of 1,000 mg/m2 immediately after the completion of nab-paclitaxel administration as part of SoC. Gemcitabine is administered on Day 1, Day 8 and Day 15 of each 28-day cycles.
Genetic: VCN-01 — VCN-01 administrated as a single IV infusion at dose 1xE13 viral particles (vp) on Day 1 of the 1st cycle and then again on Day 1 of the 4th cycle (Day 92). On cycle 1 and cycle 4, nab-paclitaxel and gemcitabine administered on Day 8, Day 15 and Day 22.
  Arms: Arm 2 -VCN-01 + SoC

SUMMARY:
A phase IIb, open-label, randomized study of Nab-Paclitaxel and Gemcitabine and plus/minus VCN-01 in Patients with Metastatic Pancreatic Cancer

DETAILED DESCRIPTION:
Multi-center, open label, randomized, 2-parallel arm, phase IIb study of nab-paclitaxel and gemcitabine as Standard of Care (SoC) plus/minus VCN-01 in patients with metastatic pancreatic cancer. Gemcitabine and nab-paclitaxel are chemotherapy drugs approved by the FDA to treat pancreatic cancer. VCN-01 is a genetically modified adenovirus characterized by the presence of four independent genetic modifications in the backbone of the wild-type human adenovirus serotype 5 (HAd5) genome that confer tumor selective replication and antitumor activity. Approximately 92 patients in sites in North America and European Union (EU) will be recruited and randomized in a 1:1 ratio to one of two treatment arms (i.e., approximately 46 patients per treatment arm):

* Arm 1- (SoC): Nab-paclitaxel and gemcitabine as SoC (28-day cycles). Patients in this arm will not receive the investigational medicinal product (IMP) VCN-01.
* Arm 2- (VCN-01+ SoC): A maximum of two (2) doses of VCN-01 administrated in combination with nab-paclitaxel and gemcitabine as SoC (28-day cycles with exception of the IMP dose cycles, which will be 35-day cycles).

A Data Monitoring Committee (DMC) will be convened at regular intervals to assess safety and to look at OS to determine if the trial can continue.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-specific procedures or assessments.
2. Male/female patients aged 18 years or over.
3. Patients with histologically or cytologically confirmed, first line metastatic pancreatic adenocarcinoma stage IV de novo, who never received previous systemic treatment for their pancreatic cancer for which the established therapy is nab-paclitaxel/gemcitabine (clinical SoC). All patients must have at least one measurable tumor lesion that can be imaged for assessments determined by RECIST 1.1.
4. Patients willing to comply with the study treatment.
5. Patients with a minimum life expectancy of 5 months.
6. ECOG performance status of 0 or 1.
7. Use of a reliable method of contraception in fertile men and women. Female patients of childbearing potential (i.e., female patients who are not postmenopausal or surgically sterile) must agree to use effective contraception. Male patients must agree to use effective contraception or be surgically sterile. All male patients must use a male condom.
8. Adequate baseline organ function (hematologic, liver, renal and nutritional)verified by laboratory analyses performed within 72 hours prior to dosing*:

   Hematology:

   • Absolute neutrophil count ≥1.5xE9 /L

   • Hemoglobin ≥9 g/dL
   * Platelets ≥100xE9/L

   Coagulation (*except in patients on anticoagulants):
   * Prothrombin time or international normalized ratio ≤1x upper limit of normal (ULN)
   * Activated partial thromboplastin time ≤1.2xULN

   Hepatic:

   • Total bilirubin ≤1.5xULN
   * ALT and AST ≤2.5xULN (if there are no liver metastases)
   * ALT and AST <5xULN, and bilirubin <1.5xULN (if there are liver metastases)

   Renal:
   * Serum creatinine ≤1.5xULN, and if >1.5xULN: Estimated creatinine clearance >50 mL/min using Cockcroft and Gault formula

   Nutritional:

   • Serum Albumin ≥30 g/L
   * Note: Adequate organ function specified in this criterion must also be met prior to VCN-01 dosing on Cycle 4 Day 1 for ARM II.

   Exclusion Criteria:

<!-- -->

1. Patients not willing to complete the study procedures for geographic, psychiatric, or social reasons.
2. Active infection or other serious illness or autoimmune disease at the moment of randomization. Active infection includes tuberculosis (TB; clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), Hepatitis B Virus (HBV; positive HBV surface antigen [HBsAg] result), Hepatitis C Virus (HCV; positive HCV Ribonucleic acid [RNA]), or human immunodeficiency virus (positive HIV 1/2 antibodies). HBV carriers (patients positive for HBsAg) or those patients requiring antiviral therapy treatment for HBV virus or HCV are not eligible to participate.

   However, the following patients are eligible to participate in the study:

   o Patients with past or resolved TB are eligible;

   o Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible. Blood HBV DNA must be obtained and must be negative in these patients prior to treatment;

   o Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
3. Treatment with live attenuated vaccines in the last 3 weeks and with the adenovirus type-5 (Ad5)-based COVID-vaccine in the last 12 weeks before the administration of study treatment.
4. Known chronic liver disease (liver cirrhosis, chronic hepatitis). If there is a suspicion of hepatic fibrosis, a FibroScan must be performed; patients with a value ≥9.5 kPa will be excluded. Note: Transient elastography (Fibroscan) is a non-invasive method for the assessment of hepatic fibrosis.
5. Treatment with another investigational agent within five of that treatment's half-lives prior to infusion of study treatment.
6. Viral syndrome diagnosed during the 2 weeks before start of study treatment administration.
7. Chronic immunosuppressive therapy and/or disease modifying therapy, except inhaled corticosteroids, and oral or IV corticosteroids with a dose lower than 10 mg prednisone or equivalent/day (exception: dexamethasone 1 mg/day as maximum).
8. Concurrent malignant hematologic or solid disease. Patients with a prior history of cancer can be allowed if complete remission for at least 3 years.
9. Patients in close contact (e.g., living in same house) with immunosuppressed patients (i.e., patients with chronic immunosuppressive therapy including high dose of corticosteroids, patients with acquired immunodeficiency syndrome (AIDS), and other chronic immune system diseases).
10. Patients with Li Fraumeni syndrome or with previously known retinoblastoma protein pathway germline deficiency.
11. A female patient, who is pregnant or lactating.
12. Patients receiving full-dose anticoagulant therapy or in whom these therapies cannot be withdrawn 2 days prior and 2 days after VCN-01 administration. Patients with uncontrolled coagulopathy should be excluded.
13. Untreated brain metastases and/or leptomeningeal carcinomatosis with progressive symptoms despite corticosteroid coverage. Patients with brain metastases with stable symptoms can be included.
14. Any other condition, disease, metabolic dysfunction (e.g., uncontrolled diabetes mellitus), active or uncontrolled infection/inflammation, physical examination finding, mental state or clinical laboratory finding that would contraindicate participation in the clinical study due to safety concerns or compliance with clinical study procedures.
15. Patients with previous pneumonitis or interstitial lung disease.
16. Patients with pre-existing sensory neuropathy >G1.
17. Patients with known risk factors for bowel perforation.
18. Patients with QT interval corrected by Fridericia (QTcF) assessment >450 ms for men or >470 ms for women and left ventricular ejection fraction (LVEF) evaluation less than 50% measured by ECHO or multigated acquisition scan.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Subjects, for whom first line treatment options other than the combination Gemcitabine/Nab-Paclitaxel are recommended by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From randomization until death for any cause up to 3 years
  Time from randomization until death in both arms
Incidence of Adverse Events after VCN-01 IV administration | From randomization until disease progression assessed up to 3 years
  Safety and tolerability of VCN-01, IV administered at Week 1 and Week 14 in Arm 2 measured as incidence of Adverse Events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Time to progression (TTP) or Progression Free Survival (PFS) | TTP: From randomization until disease progression assessed up to 3 years or death due to progression.PFS: From randomization to either progression or death from any cause.
Overall Response Rate (ORR) | From randomization until death for any cause up to 3 years
  Objective response rate (ORR) defined as the sum of patients who achieved partial response (PR) plus patients who achieved complete response (CR) using RECIST version 1.1 criteria.
Disease Control Rate (DCR) | From randomization until death for any cause up to 3 years
  Disease Control Rate (DCR) defined as: stable disease (SD) + partial response (PR) + complete response (CR)
Landmark 1-year survival | From randomization to 1-year landmark
Progression Free Survival (PFS) at the 1-year landmark | From randomization to1-year landmark
  Time from randomization to either progression or death from any cause.
Duration of Response (DoR) | From randomization to disease progression assessed up to 3 years
  Time from the date of first documented response until date of documented disease progression or death in the absence of disease progression.
Changes in tumor marker Ca 19.9 | From randomization until disease progression assessed up to 3 years
  Tumor marker Ca 19.9 measured every 4 weeks while on study

OTHER OUTCOMES:
Neutralizing anti-VCN-01 antibodies (Anti-Ad-Nabs) | From pre-dose up to 3 years
  Determination of neutralizing anti-VCN-01 antibodies (Anti-Ad-Nabs) in serum of Arm 2 patients at different time-points during the study.
  Cycle 1 (VCN-01+SoC dosing): Pre-dose on day 1, day 8, and day 15; Cycle 2 (SoC dosing): Day 1; Cycle 3 (SoC dosing): Day 1; Cycle 4 (VCN-01+SoC dosing): Pre-dose on day 1, day 8, and day 15; On Day 1 of any subsequent SoC cycle.
PH20 levels in serum | From pre-dose to end of treatment defined as 1 month after the last dose of nab-paclitaxel/gemcitabine.
  Determination of PH20 levels in serum of Arm 2 (VCN-01 + SoC) patients at the following time-points:
  Cycle 1 (VCN-01+SoC dosing): Pre-dose on day 1, 48h post-dose and on day 8; Cycle 2 (SoC dosing): Day 1; Cycle 3 (SoC dosing): Day 1; Cycle 4 (VCN-01+SoC dosing): Pre-dose on day, 48h post-dose and on day 8; On Day 1 of any subsequent SoC cycle.
VCN-01 genomes levels in blood | From pre-dose to end of treatment defined as 1 month after the last dose of nab-paclitaxel/gemcitabine.
  Determination of VCN-01 genomes in whole blood of Arm 2 (VCN-01 + SoC) patients at the following time-points:
  Cycle 1 (VCN-01+SoC dosing): Pre-dose and 4h post-dose on day 1, 48h post-dose, on day 8 and day 15; Cycle 2 (SoC dosing): Day 1; Cycle 3 (SoC dosing): Day 1; Cycle 4 (VCN-01+SoC dosing): Pre-dose and 4h post dose on day 1, 48h post-dose, on day 8 and day 15; On Day 1 of any subsequent SoC cycle.
Immune markers | From pre-dose to end of treatment defined as 1 month after the last dose of nab-paclitaxel/gemcitabine.
  Determination of immune markers in serum of Arm 1 (SoC) or Arm 2 (VCN-01 + SoC) patients at the following time-points:
  Arm 1:
  Cycle 1 (SoC): Pre-dose on day 1, day 8 and day 15. On Day 1 of any subsequent SoC cycle.
  Arm 2:
  Cycle 1 (VCN-01+SoC dosing): Pre-dose, 4h and 48h post-dose and on day 8; Cycle 2 (SoC dosing): Day 1; Cycle 3 (SoC dosing): Day 1; Cycle 4 (VCN-01+SoC dosing): Pre-dose, 4h and 48h post-dose, on day 8 and day 15; On Day 1 of any subsequent SoC cycle.
Radiomics | Changes from baseline to every 8 week or every 4 weeks if there is a suspicion of Progressive Disease (PD) not radiologically confirmed during treatment and until disease progression up to 3 years.
  Change in radiomics assessed from the images of CT scans or MRI.
Tumor growth | Changes from baseline to every 8 week or every 4 weeks if there is a suspicion of Progressive Disease (PD) not radiologically confirmed during treatment and until disease progression up to 3 years.
  Change in tumor growth assessed from the images of CT scans or MRI.
Changes in Quality of Life (QoL) via the validated Quality of Life Questionnaire of the European Organization for Research and Treatment of Cancer (EORTC QLQ-C30) version 3. | From Day 1 in first treatment cycle (35-days) to last follow-up visit up to 3 years.
  Changes in QoL assessed as the difference between QoL in day 1 of 1st treatment cycle (35 d) to QoL in day 1 of Cycle 2 (28d), to QoL in day 1 of Cycle 3 (28d), to QoL in day 1 of Cycle 4 (35d) and to QoL in day 1 of any subsequent SoC cycle (28d).
  Changes in QoL in EoT visit (1 month after last SoC treatment).
  Changes in QoL until disease progression in each monthly follow-up visit.
  After disease progression, changes in QoL in each monthly follow up visit during the first 6 months; changes in bimonthly follow-up visits up to to 2 years from progression and changes in each follow-up visit every 6 months onwards.
  The QoL scale ranges in score from 0 to 100, a high score represents a higher response level.
Disease Control Rate (DCR) to subsequent therapies | From disease progression to exitus for any cause up to 3 years
  Disease Control Rate (DCR) defined as: stable disease (SD) + partial response (PR) + complete response (CR)

CONTACTS AND LOCATIONS:
Overall Officials: Tara E Seery, MD, Principal Investigator — Hoag Memorial Hospital Presbyterian; Edward Kim, MD, PhD, Principal Investigator — University of California, Davis Cancer Centre; Vivek R Sharma, MD, FACP, Principal Investigator — University of Louisville, Brown Cancer Center; Alana TH Nguyen, MD, PhD, Principal Investigator — Weill Medical College of Cornell University; Arjun Mittra, MD, Principal Investigator — Martha Morehouse Tower; Christopher Nevala-Plagemann, MD, Principal Investigator — Hunstman Cancer Institute, University of Utah; Alexander Spira, MD, PhD, Principal Investigator — Virginia Cancer Specialists; Rocío García, MD, PhD, Principal Investigator — Hospital Universtario 12 de octubre; Teresa Macarulla, Md, PhD, Principal Investigator — Hospital Vall d'Hebron; Andrés Muñoz, MD, PhD, Principal Investigator — Hospital Gregorio-Marañon; Carmen Guillén-Ponce, MD, PhD, Principal Investigator — Hospital Universitario Ramon y Cajal; Miriam Lobo, MD, PhD, Principal Investigator — Hospital General Universitario de Valencia; Roberto Pazo, MD, PhD, Principal Investigator — Hospital Miguel Servet; Inmaculada Gallego, MD, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío; Berta Laquente, MD. PhD, Principal Investigator — Hospital Duran i Reynals (ICO); Eva Martinez de Castro, MD, PhD, Principal Investigator — Hospital Universitario Marqués de Valdecilla; Mireya Cazorla, MD, PhD, Principal Investigator — Hospital Universitario Virgen de la Victoria
Locations (17):
- United States (7):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California - Davis Cancer Center, Sacramento, California
  - University of Louisville - Brown Cancer Center, Louisville, Kentucky
  - Weill Cornell Medical Center, New York, New York
  - Martha Morehouse Tower, Columbus, Ohio
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
- Spain (10):
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Hospital Duran i Reynals (ICO), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Gregorio Marañon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Univesitario de Valencia, Valencia
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No